CLINICAL TRIAL: NCT02251847
Title: The Efficacy and Safety of a Combination Therapy of Rosuvastatin and Ezetimibe Versus Monotherapy of Rosuvastatin in Hypercholesterolemia Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-ROEZ-301
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Hypercholesterolemia
Keywords: cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- R5 (Active Comparator): Rosuvastatin 5mg
  Interventions: Drug: Rosuvastatin/Ezetimibe
- R10 (Active Comparator): Rosuvastatin 10mg
  Interventions: Drug: Rosuvastatin/Ezetimibe
- R20 (Active Comparator): Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin/Ezetimibe
- R5/E10 (Experimental): Rosuvastatin 5mg/ezetimibe 10mg
  Interventions: Drug: Rosuvastatin/Ezetimibe
- R10/E10 (Experimental): Rosuvastatin 10mg/ezetimibe 10mg
  Interventions: Drug: Rosuvastatin/Ezetimibe
- R20/E10 (Experimental): Rosuvastatin 20mg/ezetimibe 10mg
  Interventions: Drug: Rosuvastatin/Ezetimibe

INTERVENTIONS:
Drug: Rosuvastatin/Ezetimibe — Rosuvastatin 5mg

SUMMARY:
To evaluate efficacy and safety of a combination therapy of rosuvastatin and ezetimibe versus monotherapy of rosuvastatin in hypercholesterolemia patients

DETAILED DESCRIPTION:
To evaluate efficacy and safety of a combination therapy of rosuvastatin and ezetimibe versus monotherapy of rosuvastatin in hypercholesterolemia patients

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemic patient

Exclusion Criteria:

* Has history of hypersensitivity to HMG-CoA reductase inhibitor and Ezetimibe

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline to 8 week in LDL-Cholesterol | baseline and 8 week

SECONDARY OUTCOMES:
Percent change from baseline to 4 week in LDL-Cholesterol | baseline and 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hoon Ahn, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gil Medical Center, Seoul, South Korea